CLINICAL TRIAL: NCT06167694
Title: A Multicenter, Open Phase Ib/II Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of HRS-8080 in Combination With Dalpiciclib Isethionate Tablets in Patients With ER-positive, HER2-negative Unresectable or Metastatic Breast Cancer
Brief Title: Clinical Study of HRS-8080 in Combination With Dalpiciclib Isethionate Tablets in Patients With Unresectable or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-201
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Unresectable or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Multi-center, open clinical study of HRS-8080 in conjunction with Dalpiciclib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group A (Experimental)
  Interventions: Drug: HRS-8080; Dalpiciclib Isethionate Tablets

INTERVENTIONS:
Drug: HRS-8080; Dalpiciclib Isethionate Tablets — HRS-8080 combined with Dalpiciclib Isethionate Tablets

SUMMARY:
This is a multicenter, open phase Ib/II clinical study, which is divided into two phases: dose exploration and efficacy expansion. Participants entering the study will receive HRS-8080 combined with Dalpiciclib Isethionate Tablets therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-75 years with both ends included.
2. ECOG Physical status 0-1 points.
3. Patients with histologically confirmed metastatic or locally advanced breast cancer.
4. Dose-exploration stage: advanced stage has received at least 1 line of endocrine therapy progression in the past, efficacy extension stage: has not received any systemic treatment for advanced disease5.
5. Antitumor therapy with radiographically confirmed disease progression or receiving advanced first-line standard endocrine therapy with no clinical or radiographically confirmed disease progression.
6. At least one measurable extracranial lesion must be present.
7. Expected survival >3 months.
8. The functional level of the organ must meet the requirements of the test.
9. Fertile female subjects must consent to use highly effective contraception during the study treatment period and for 7 months after the end of the study treatment period; Fertile female subjects must be negative for serum HCG within 7 days prior to study enrollment and must be non-lactating.
10. Volunteer to participate in this clinical trial, be willing and able to follow clinical visit and study related procedures, understand study procedures and have signed informed consent.

Exclusion Criteria:

1. Symptoms of visceral metastasis.
2. Previous treatment did not meet trial requirements.
3. Received nitrosourea or mitomycin within 6 weeks before the first dose in this study; Received major organ surgery, cytotoxic drugs, immunotherapy, targeted therapy, anti-tumor traditional Chinese medicine or other clinical investigational drugs within 4 weeks before the first medication; He received endocrine therapy and palliative radiotherapy within 2 weeks before the first dose.
4. Less than 14 days after the first dose of CYP3A4; CYP3A4 is treated with a strong inducer <28 days from the date of first administration.
5. Patients with active (untreated or clinically symptomatic) brain metastases, cancerous meningitis, spinal cord compression, or a history of primary tumors of the central nervous system.
6. A history of clinically severe cardiovascular disease.
7. Patients with uncontrolled tumor-related pain as judged by the investigator.
8. Those who received immunosuppressive agents or systemic hormone therapy for immunosuppression within 2 weeks prior to the first dose.
9. The damage caused by the subject receiving other treatments has been recovered.
10. Severe infection occurred within 4 weeks prior to the second dose.
11. The first study investigated the occurrence of arteriovenous thrombosis within 6 months prior to medication.
12. Patients with clinically significant endometrial abnormalities.
13. Untreated active hepatitis.
14. Subjects had other malignancies within the past 5 years or currently.
15. Have an inherited or acquired bleeding tendency.
16. History of active autoimmune disease, immune deficiency, and autoimmune disease.
17. One of the many factors that affect oral medications.
18. Subjects are acutely infected or have active TB and require medication.
19. Known allergy to HRS-8080 ingredient, Dalpiciclib and ingredient.
20. Pregnant and lactating women or women planning to become pregnant during the study period.
21. There is a clear history of neurological or psychiatric disorders and the subjects have a history of psychotropic substance abuse or drug use.
22. The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participating in the study or interfere with the study results, as well as patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | About 2 years
Maximum tolerated dose (MTD) | About 2 years
Recommended phase II dose (RP2D) | About 2 years
Safety endpoints: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | About 2 years
Outcome endpoint: Objective Response Rate (ORR) | About 2 years

SECONDARY OUTCOMES:
Steady-state peak concentration (Cmax,ss) | About 2 years
Steady-state peak time (Tmax,ss) | About 2 years
Steady-state valley concentration (Cmin,ss) | About 2 years
Steady-state blood drug concentration-time curve area (AUCss) | About 2 years
Best overall response (BOR) | About 2 years
Duration of response (DoR) | About 2 years
Disease control rate (DCR) | About 2 years
Clinical benefit rate (CBR) | About 2 years
Progression-free survival (PFS) | About 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese PLA General Hospital Fifth Medical Center, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided